CLINICAL TRIAL: NCT02912182
Title: Acute Unilateral Vestibulopathy and Corticosteroid Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Placebo medication expired
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VN-FT-01
Record Dates: First submitted 2016-09-15; First posted 2016-09-23 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Vestibular Diseases; Vestibular Neuronitis
MeSH Terms: conditions — Vestibular Diseases; Vestibular Neuronitis | interventions — Betamethasone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Day 1: Intravenous sodium-chloride 2ml Day 2-6: 10 tablets placebo Day 7: 8 tablets placebo Day 8: 6 tablets placebo Day 9: 4 tablets placebo Day 10: 2 tablets placebo Day 11: 1 tablet placebo
  Interventions: Drug: Placebo
- Short treatment (Active Comparator): Day 1: Intravenous betamethasone 8mg (2ml of 4mg/ml) Day 2-3: 10 tablets prednisolone 5 mg Day 4-6: 10 tablets placebo Day 7: 8 tablets placebo Day 8: 6 tablets placebo Day 9: 4 tablets placebo Day 10: 2 tablets placebo Day 11: 1 tablet placebo
  Interventions: Drug: Betamethasone; Drug: Prednisolone
- Standard treatment (Active Comparator): Day 1: Intravenous betamethasone 8mg (2ml of 4mg/ml) Day 2-6: 10 tablets prednisolone 5 mg Day 7: 8 tablets prednisolone 5 mg Day 8: 6 tablets prednisolone 5 mg Day 9: 4 tablets prednisolone 5 mg Day 10: 2 tablets prednisolone 5 mg Day 11: 1 tablet prednisolone 5 mg
  Interventions: Drug: Betamethasone; Drug: Prednisolone

INTERVENTIONS:
Drug: Betamethasone — Betamethasone intravenous
  Other Names: Betapred
  Arms: Short treatment; Standard treatment
Drug: Placebo — Placebo intravenous NaCl intravenous administration Placebo tablets
  Other Names: Sodiumchloride
  Arms: Placebo
Drug: Prednisolone — Oral tablets
  Other Names: Prednisolon
  Arms: Short treatment; Standard treatment

SUMMARY:
Randomized placebo controlled trial on patients suffering from acute unilateral vestibulopathy. Patients will be randomized into 3 arms; 1) Placebo only, 2) Short corticosteroid treatment (3days) 3) Longer corticosteroid treatment (11 days).

Vestibular function as well as subjective symptoms will be estimated in the acute stage and regularly up to one year after the debut.

DETAILED DESCRIPTION:
Randomized controlled trial in 3 arms to see if a short or a even shorter period of steroid treatment on patients diagnosed with vestibular neuritis can be as effective as the only comparable study thus far (Strupp et al, NEJM 22, 351(4) 354-61). If a shorter treatment with a lower dose has the same outcome, then more patients might be eligible for the treatment as many are excluded due to risk for adverse effects.

Corticosteroid treatment in acute unilateral vestibulopathy has recently been the subject for a Cochrane review with the conclusion of insufficient evidence for treatment effect and recommend studies with subjective symptom based evaluation together with functional testing.

Patients with acute unilateral vestibulopathy diagnosed within 48hrs after debut. The patients (after acceptance) will be randomized into either of 3 arms and will receive placebo/short treatment (3days)/standard treatment (in Sweden 11 days).

Patients will record subjective symptoms according to Liknert scale during the acute stage and fill out enquiries after 3 and 12 months.

Vestibular function will be assessed with caloric irrigation and video-Head-Impulse-Test (vHIT) as soon as possible after the debut and again after 1, 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* definite unilateral vestibulopathy
* no pathological HINTS (examination criteria in acute vestibular syndrome)
* capable of making their own decisions

Exclusion Criteria:

* tinnitus or hearing loss with same debut as vertigo
* history of bleeding peptic ulcer
* glaucoma
* pregnancy or non-acceptance to use anticonception measures during 13 days after debut
* high blood pressure >180 systolic, 105, diastolic
* ketoacidosis with a Base Excess >=2
* psychic disorder (not including mild depression)
* serious infection (neutropenia, tuberculosis)
* chronic otitis
* history of vertiginous disease; Ménière, Vertiginous migraine, atypical BPPV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-12; Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Caloric function | after 3 months
  Warm (44deg C) and cold (30 deg C) water irrigation of the ear canals of both ears. Jongkees formula (ratio of response between the ears) is assessed for abnormal or normal function
Caloric function | 1 year
  Warm (44deg C) and cold (30 deg C) water irrigation of the ear canals of both ears. Jongkees formula (ratio of response between the ears) is assessed for abnormal or normal function

SECONDARY OUTCOMES:
vHIT | 2-5 days after debut
  measurement of vestibulo-ocular reflex in all semicircular canals. Gain <0.7 (ratio between head and eye movement) is regarded as pathological
Subjective visual vertical/horizontal | 2-5 days after debut,
  Assessment of spatial orientation or utricular function (of the inner ear) as a measure of degree of vestibular loss and of compensation
Covert saccades | 2-5 days after debut,
  Covert catch-up eye saccades are sometimes seen during vHIT. The origin is unknown. The frequency as well as latency times will be analyzed and correlated to subjective measures
Vertigo Diary | Daily from debut and until no subjective vertigo is experienced, longest 4 weeks
  Self-assessment of vertigo according to a Liknert scale daily (1= no vertigo and 10= worst possible vertigo
Sleep Diary | Daily from debut and 14 days onwards (2 days after last treatment)
  Patients often experience troubled sleep when treated with corticosteroids. How much has not been assessed. The patients will assess their sleep the previous night according to a Liknert scale (1=good nights sleep, 10=hardly slept at all)
HADS-enquiry | 3 and 12 months after debut
  Hospital Anxiety and Depression Scale. To asses the degree of anxiety and depression among the patients, often associated with chronic dizziness
VSS-enquiry | 3 and 12 months after debut
  Vertigo sympton score, To assess vertigo symptoms
DHI-enquiry | 3 and 12 months after debut
  Dizziness Handicap Inventory, to assess the degree of how dizziness affect daily life
VHQ-enquiry | 3 and 12 months after debut
  Vertigo Handicap Questionnaire. To assess the degree of how vertigo affect daily life
Stress hormones | At debut and 1 year
  Measurement of Plasma thyroid hormones, adrenocorticoid hormones (ACTH, Cortisone) as stress indicators in acute vertigo. Baseline will be taken 1 year after debut
Saliva-Cortisol | At debut and up to 1 week
  Daily measurement of saliva cortisol as measurement of stress
Adverse Events | From debut to 1 year after
  Analysis of adverse events to treatment as well as functional outcome
Hospital stay | From debut up to 10 days
  Duration of hospital stay
vHIT | 1 year
  measurement of vestibulo-ocular reflex in all semicircular canals. Gain <0.7 (ratio between head and eye movement) is regarded as pathological
Subjective visual vertical/horizontal | 1 month
  Assessment of spatial orientation or utricular function (of the inner ear) as a measure of degree of vestibular loss and of compensation
Subjective visual vertical/horizontal | 3 months
  Assessment of spatial orientation or utricular function (of the inner ear) as a measure of degree of vestibular loss and of compensation
Subjective visual vertical/horizontal | 1 year
  Assessment of spatial orientation or utricular function (of the inner ear) as a measure of degree of vestibular loss and of compensation
Covert saccades | 3 months
  Covert catch-up eye saccades are sometimes seen during vHIT. The origin is unknown. The frequency as well as latency times will be analyzed and correlated to subjective measures
Covert saccades | 1 year
  Covert catch-up eye saccades are sometimes seen during vHIT. The origin is unknown. The frequency as well as latency times will be analyzed and correlated to subjective measures
Sick-leave | debut up to 1 year
  Time needed for sick-leave
Daily living | debut up to 1 year
  Time until daily activities are as prior to th disease

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Tjernström, MD, PhD, Principal Investigator — Lund University
Locations (3):
- Sweden (3):
  - Dept OtoRhinoLaryngology, Helsingborg
  - Dept. Otorhinolaryngology, Kristianstad
  - Dept. OtoRhinoLaryngology Head and Neck Surgery, Skane University Hospital, Lund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fishman JM, Burgess C, Waddell A. Corticosteroids for the treatment of idiopathic acute vestibular dysfunction (vestibular neuritis). Cochrane Database Syst Rev. 2011 May 11;2011(5):CD008607. doi: 10.1002/14651858.CD008607.pub2. PMID 21563170
- [Result] Strupp M, Zingler VC, Arbusow V, Niklas D, Maag KP, Dieterich M, Bense S, Theil D, Jahn K, Brandt T. Methylprednisolone, valacyclovir, or the combination for vestibular neuritis. N Engl J Med. 2004 Jul 22;351(4):354-61. doi: 10.1056/NEJMoa033280. PMID 15269315